CLINICAL TRIAL: NCT03080402
Title: Mechanical Perturbation Training for ACL Injury Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Delaware (Other)
Collaborators: Simbex, LLC (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lynn Snyder-Mackler, Alumni Distinguished Professor, University of Delaware
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R44HD068054 (NIH); 5R44HD068054 (NIH)
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Anterior Cruciate Ligament Injury; ACL
Keywords: Anterior Cruciate Ligament; ACL injury; Injury prevention; Perturbation training; Risk factors
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: 24 female athletes (12 with high KAM; 12 with normal KAM) will be recruited into the intervention/ testing phase of this study. Female athletes with KAM > 25.25 Nm will be classified as high KAM and will receive 12 sessions of mechanically-driven perturbation training and female athletes with KAM < 25.25 Nm will be classified as normal KAM and only participate in baseline performance testing, followed 6 weeks later by another session of drop jump motion analysis and performance testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High KAM (Experimental): Mechanically-driven neuromuscular training. 2 times per week for 6 weeks for a total of 12 sessions. Perturbation training
  Interventions: Device: Mechanical Perturbation Training
- Normal KAM (No Intervention): No intervention

INTERVENTIONS:
Device: Mechanical Perturbation Training — The training program will consist of three stages and subjects will progress through each neuromuscular training stage.The training will consist of double- to single-limb movements with progression of jumping, hopping, and pivoting maneuvers on the perturbation device with an emphasis on proper technique and landing. The initial four sessions will focus on primarily on jumping and hopping maneuvers on double- and single-limb in the sagittal plane. The intermediate four sessions will incorporate additional medial and lateral maneuvers with the plyometric tasks. The final four sessions will incorporate rotational and pivoting activities with the maneuvers. The resultant protocol has been derived and optimized from previous published research studies and prevention techniques.
  Other Names: Reactive Agility Platform Trainer 2.0; RAPTr
  Arms: High KAM

SUMMARY:
A prospective trial will be used to evaluate the efficacy of prophylactic mechanical perturbation training program. 24 female athletes who are regular participants in activities that involve cutting, pivoting, jumping, and lateral movements prior to injury who range in age from 15-30 year are eligible. Using a prospective risk stratification design, female athletes with knee abduction moment (KAM) > 25.25 Nm from drop jump motion analysis will be classified as high KAM and will receive 12 sessions of mechanically-driven perturbation training and female athletes with KAM < 25.25 Nm from drop jump motion analysis will be classified as normal KAM and only participate in baseline performance testing, followed 6 weeks later by another session of drop jump motion analysis and performance testing.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injuries are prevalent in sports with female athletes at particularly high risk. Female athletes have 2-4x higher risk of ACL injury compared to their male counterparts in the same high-risk sports. Modifiable and non-modifiable risk factors play a role in the high incidence of ACL injuries in female athletes. High knee abduction moment (KAM), is a known modifiable risk factor for ACL injury risk. Female athletes with a KAM greater than 25.25 Nm have been identified as at high risk for an ACL injury. The ability to classify female athletes who are at a high risk for an ACL injury, highlights the importance of identifying modifiable risk factors that can be readily addressed by physical therapists and developing targeted treatments to potentially reduce ACL injury risk while improving functional performance.

Neuromuscular training programs are treatments designed to help improve coordination, strength, and control. Such training programs have been designed to alter biomechanical and neuromuscular measures, in particular high KAM, in order to improve performance and function and thereby reduce the risk of ACL injury. Neuromuscular training programs involving plyometric exercises can reduce dynamic lower extremity valgus and limb-to-limb asymmetries in healthy female athletes. Despite the reductions in injury rates seen with performance of neuromuscular training programs, incidence of ACL injuries is remains higher than acceptable. Novel training methods are currently in development to optimize these current ACL injury prevention programs. As unanticipated perturbations may contribute to ACL injury risk, incorporating a mechanical platform device that provides unanticipated surface compliance changes (i.e. the floor lowering down below a subject's feet) into an ACL injury prevention program has the potential to optimize knee biomechanics and neuromuscular performance, including during unanticipated perturbations.

Mechanical perturbation has been advocated for as an effective training method to modify the sensorimotor system and restore normal neuromuscular coordination through exposing the subjects to controlled, progressive perturbations. Furthermore, mechanical perturbation has the potential to improve dynamic postural stability and control, and enhance muscle activation patterns. One advantage of mechanical perturbation devices is that they can be utilized while performing a variety of dynamic tasks such as hopping and jumping compared to static loading tasks such as standing and balancing activities. Dynamic tasks may place a greater demand on the knee joint, promoting joint stability as the subject overcomes the perturbation. Additionally, mechanical perturbation may allow physical therapists to administer random perturbations at different phases of the activities (i.e. as the subject is landing from a hop, or taking-off from a jump) that simulate real-life perturbations which occur during different functional or sporting activities.

The goal of this study is to assess the effectiveness of an intensive neuromuscular training program to reduce risk factors associated with ACL injury

ELIGIBILITY:
Inclusion Criteria:

* Female athletes will be eligible if they are: 1) regular participants in Level 1 and 2 sports (cutting and pivoting type sports, and 2) ages 15-30 years

Exclusion Criteria:

* History of major injury or surgery to the legs.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak knee abduction moment | baseline and 6 weeks after baseline testing
  Peak knee abduction moment during a drop jump landing task as assessed via motion analysis

SECONDARY OUTCOMES:
Peak Quadriceps torque 60 degrees/sec | baseline and 6 weeks after baseline testing
  Peak Quadriceps torque 60 degrees/sec
Peak Quadriceps torque 240 degrees/sec | baseline and 6 weeks after baseline testing
  Peak Quadriceps torque 240 degrees/sec
Peak Hamstrings torque 60 degrees/sec | baseline and 6 weeks after baseline testing
  Peak Hamstrings torque 60 degrees/sec
Peak Hamstrings torque 240 degrees/sec | baseline and 6 weeks after baseline testing
  Peak Hamstrings torque 240 degrees/sec
Single hop for distance LSI | baseline and 6 weeks after baseline testing
  Single hop for distance limb symmetry index
Crossover hop for distance LSI | baseline and 6 weeks after baseline testing
  Crossover hop for distance limb symmetry index
Triple hop for distance LSI | baseline and 6 weeks after baseline testing
  Triple hop for distance limb symmetry index
6m Timed Hop LSI | baseline and 6 weeks after baseline testing
  6 meter Timed Hop limb symmetry index

OTHER OUTCOMES:
Vertical Jump | baseline and 6 weeks after baseline testing
  Vertical jump for height

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Snyder-Mackler, PT, ATC, ScD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Physical Therapy Department, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no IPD sharing plan.